CLINICAL TRIAL: NCT05099419
Title: Motor Cortical Neuromodulation With Repetitive Transcranial Magnetic Stimulation in Women With Overactive Bladder and Urgency Urinary Incontinence
Brief Title: Repetitive Transcranial Magnetic Stimulation in Women With Overactive Bladder With Urgency Incontinence
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Larissa Rodriguez, Professor of Urology, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HS-21-00578
Record Dates: First submitted 2021-09-29; First posted 2021-10-29 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Overactive Bladder; Urge Incontinence
Keywords: Repetitive Transcranial Magnetic Stimulation; Overactive Bladder; Urge Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Two different intervention protocols will be administered in a crossover design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- High Frequency rTMS Protocol (Experimental): High frequency with 10 Hz at 80% motor threshold intensity with figure-of-eight coil for a total of 2,000 pulses. Pulses will be delivered in 10-second trains with a 50-second pause between the trains.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Low Frequency rTMS Protocol (Experimental): Low frequency 1 Hz at 80% motor threshold intensity with figure-of-eight coil for a total of 2,000 pulses. Pulses will be delivered continuously.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — rTMS uses pulses of magnetic energy to non-invasively stimulate the brain. The rTMS device to be used in this study is the Magstim Rapid2 Plus1. The rTMS device is connected to an active figure-of-eight coil which rests against the scalp and delivers the magnetic energy to the brain. The rTMS protocol is specified by the parameters of pulse frequency, duration of continuous pulse delivery, intensity, and stimulation location.
  Each participant will receive two different standard rTMS protocols that have been used in past research studies for modulation of pelvic floor tone delivered over the motor cortex in an area that is known to control pelvic floor muscles.

SUMMARY:
Overactive bladder (OAB) affects an estimated 16-30% of women in the US and urgency urinary incontinence (UUI) affects 7-11% of women with OAB. It is known that repetitive transcranial magnetic stimulation (rTMS) over the supplementary motor area (SMA) can modulate the pelvic floor muscle activity with potential benefits for various urologic conditions. The goal of this study is to assess feasibility of rTMS as a treatment option for OAB with UUI by determining which rTMS frequency is most effective in targeting sensory components of OAB, namely urinary urgency, and also in targeting the brain network known to be involved in OAB.

DETAILED DESCRIPTION:
Eligible participants with OAB and UUI will undergo resting state functional MRI of the brain to map baseline brain activity. Participants will then undergo rTMS of the SMA with electromyography (EMG) monitoring of the pelvic floor muscles. They will then undergo another MRI to assess and changes in brain activity due to rTMS. Participants will be asked about their bladder symptoms over the course of the study.

The study will have a crossover design. The investigators plan to recruit 10 women with symptoms of OAB and UUI. During the first week, participants will be screened, asked to fill out a bladder questionnaire, and to complete a bladder diary. During the next two weeks, participants will undergo rTMS and functional MRI of the brain to assess brain activity.

All participants will undergo two different known rTMS protocols for the pelvic floor, high-frequency and low-frequency, separated by a 1-week washout period. Each participant will be randomized to which protocol they will have first. In total, 5 participants will have started with high-frequency rTMS first and 5 participants will have started with low-frequency rTMS. At the end, all participants will have undergone both high- and low-frequency rTMS.

The primary objective of the study is to assess the feasibility of rTMS in patients with OAB and UUI, which will be assessed with recruitment and retention rates of participants. The investigators also aim to determine if SMA activity mediates OAB symptoms and pelvic floor muscle tone using functional MRI of the brain. Finally, the investigators want to assess bladder symptoms following rTMS using participant questionnaires and number of UUI episodes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* female
* diagnosis of overactive bladder with symptoms of urgency urinary incontinence majority of the time during the last 3 months

Exclusion Criteria:

* current use of sacral neuromodulation
* new initiation of overactive bladder treatment within the last 6 weeks
* has had intradetrusor onabotulinumtoxinA injections in the last 3 months
* neurological disease affecting the bladder or bowel
* incomplete bladder emptying
* history of urologic cancer
* active infection
* history of cystitis caused by tuberculosis, radiation, or chemotherapies
* severe pelvic pain
* pregnancy
* post-partum 6 weeks
* post-surgical 6 weeks
* cannot undergo MRI
* history of epilepsy or seizures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Effects of repetitive transcranial magnetic stimulation (rTMS) on pelvic-supplementary motor area (SMA) activity after low-frequency rTMS | Functional MRI lasting 30 minutes will be obtained immediately before low-frequency rTMS during weeks 2 and 3.
  The effects of low-frequency rTMS on brain activity will be evaluated with functional MRI performed immediately before the rTMS session and also after 30 minutes after the session in order to document interval changes.
Effects of repetitive transcranial magnetic stimulation (rTMS) on pelvic-supplementary motor area (SMA) activity after low-frequency rTMS | Functional MRI lasting 30 minutes will be obtained within 30 minutes of finishing low-frequency rTMS during weeks 2 and 3.
  The effects of low-frequency rTMS on brain activity will be evaluated with functional MRI performed immediately before the rTMS session and also after 30 minutes after the session in order to document interval changes.
Effects of rTMS on pelvic-SMA activity after high-frequency rTMS | Functional MRI lasting 30 minutes will be obtained immediately before high-frequency rTMS during weeks 2 and 3.
  The effects of high-frequency rTMS on brain activity will be evaluated with functional MRI performed immediately before the rTMS session and also after 30 minutes after the session in order to document interval changes.
Effects of rTMS on pelvic-SMA activity after high-frequency rTMS | Functional MRI lasting 30 minutes will be obtained within 30 minutes of finishing high-frequency rTMS during weeks 2 and 3.
  The effects of high-frequency rTMS on brain activity will be evaluated with functional MRI performed immediately before the rTMS session and also after 30 minutes after the session in order to document interval changes.
Effects of rTMS on pelvic floor muscle activity after low-frequency rTMS | Pelvic floor EMG will be obtained during low-frequency rTMS session, lasting 33 minutes, during weeks 2 and 3.
  The effects of low-frequency rTMS on pelvic floor muscle activity will be evaluated with pelvic floor electromyography (EMG) obtained with a rectal sensor during the low-frequency rTMS session.
Effects of rTMS on pelvic floor muscle activity after high-frequency rTMS | Pelvic floor EMG will be obtained during high-frequency rTMS session, lasting 20 minutes, during weeks 2 and 3.
  The effects of high-frequency rTMS on pelvic floor muscle activity will be evaluated with pelvic floor electromyography (EMG) obtained with a rectal sensor during the high-frequency rTMS session.

SECONDARY OUTCOMES:
Assess subjective OAB and UUI symptom changes following rTMS | Subjective OAB and UUI symptoms will be assessed with the OAB-q at baseline during week 1.
  OAB and UUI symptoms will be assessed with the overactive bladder questionnaire (OAB-q). This validated instrument contains 33 questions regarding bladder symptoms and quality of life associated with OAB rated on a 6-point Likert scale. The total score ranges from 0 to 100 with higher scores reflecting greater degree of symptom bother.
Assess subjective OAB and UUI symptom changes following rTMS | Subjective OAB and UUI symptoms will be assessed with the OAB-q after rTMS treatments during weeks 2 and 3.
  OAB and UUI symptoms will be assessed with the overactive bladder questionnaire (OAB-q). This validated instrument contains 33 questions regarding bladder symptoms and quality of life associated with OAB rated on a 6-point Likert scale. The total score ranges from 0 to 100 with higher scores reflecting greater degree of symptom bother.
Assess objective OAB and UUI symptom changes following rTMS | Objective OAB and UUI symptoms will be assessed with a bladder diary at baseline during week 1.
  Objective OAB and UUI symptoms will be assessed with a bladder diary where participants will document number of voids, volume of voids, urgency episodes, and episodes of urgency incontinence in the past 24 hours.
Assess objective OAB and UUI symptom changes following rTMS | Objective OAB and UUI symptoms will be assessed with a bladder diary after rTMS treatments during weeks 2 and 3.
  Objective OAB and UUI symptoms will be assessed with a bladder diary where participants will document number of voids, urgency episodes, and episodes of urgency incontinence in the past 24 hours.

OTHER OUTCOMES:
Feasibility of repetitive transcranial magnetic stimulation (rTMS) use in women with overactive bladder (OAB) and urgency urinary incontinence (UUI) | Feasibility will be assessed after completion of the study, up to 6 months.
  Feasibility will be assessed with recruitment and retention rates, time required to achieve target number of eligible participants, and completion rates of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Rodriguez, MD, Study Director — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reynolds WS, Fowke J, Dmochowski R. The Burden of Overactive Bladder on US Public Health. Curr Bladder Dysfunct Rep. 2016 Mar;11(1):8-13. doi: 10.1007/s11884-016-0344-9. Epub 2016 Jan 23. PMID 27057265
- [Background] Burgio KL, Locher JL, Goode PS, Hardin JM, McDowell BJ, Dombrowski M, Candib D. Behavioral vs drug treatment for urge urinary incontinence in older women: a randomized controlled trial. JAMA. 1998 Dec 16;280(23):1995-2000. doi: 10.1001/jama.280.23.1995. PMID 9863850
- [Background] Lightner DJ, Gomelsky A, Souter L, Vasavada SP. Diagnosis and Treatment of Overactive Bladder (Non-Neurogenic) in Adults: AUA/SUFU Guideline Amendment 2019. J Urol. 2019 Sep;202(3):558-563. doi: 10.1097/JU.0000000000000309. Epub 2019 Aug 8. PMID 31039103
- [Background] Yani MS, Fenske SJ, Rodriguez LV, Kutch JJ. Motor cortical neuromodulation of pelvic floor muscle tone: Potential implications for the treatment of urologic conditions. Neurourol Urodyn. 2019 Aug;38(6):1517-1523. doi: 10.1002/nau.24014. Epub 2019 May 1. PMID 31044482
- [Background] Griffiths D. Imaging bladder sensations. Neurourol Urodyn. 2007 Oct;26(6 Suppl):899-903. doi: 10.1002/nau.20488. PMID 17654564
- [Background] Blok BF, Willemsen AT, Holstege G. A PET study on brain control of micturition in humans. Brain. 1997 Jan;120 ( Pt 1):111-21. doi: 10.1093/brain/120.1.111. PMID 9055802
- [Background] Griffiths D, Tadic SD, Schaefer W, Resnick NM. Cerebral control of the bladder in normal and urge-incontinent women. Neuroimage. 2007 Aug 1;37(1):1-7. doi: 10.1016/j.neuroimage.2007.04.061. Epub 2007 May 18. PMID 17574871
- [Background] Griffiths D, Clarkson B, Tadic SD, Resnick NM. Brain Mechanisms Underlying Urge Incontinence and its Response to Pelvic Floor Muscle Training. J Urol. 2015 Sep;194(3):708-15. doi: 10.1016/j.juro.2015.03.102. Epub 2015 Mar 28. PMID 25828973
- [Background] Tadic SD, Griffiths D, Schaefer W, Murrin A, Clarkson B, Resnick NM. Brain activity underlying impaired continence control in older women with overactive bladder. Neurourol Urodyn. 2012 Jun;31(5):652-8. doi: 10.1002/nau.21240. Epub 2012 Mar 30. PMID 22473921
- [Background] Brusa L, Finazzi Agro E, Petta F, Sciobica F, Torriero S, Lo Gerfo E, Iani C, Stanzione P, Koch G. Effects of inhibitory rTMS on bladder function in Parkinson's disease patients. Mov Disord. 2009 Feb 15;24(3):445-8. doi: 10.1002/mds.22434. PMID 19133657
- [Background] Nizard J, Esnault J, Bouche B, Suarez Moreno A, Lefaucheur JP, Nguyen JP. Long-Term Relief of Painful Bladder Syndrome by High-Intensity, Low-Frequency Repetitive Transcranial Magnetic Stimulation of the Right and Left Dorsolateral Prefrontal Cortices. Front Neurosci. 2018 Dec 11;12:925. doi: 10.3389/fnins.2018.00925. eCollection 2018. PMID 30618554
- [Background] Lefaucheur JP, Andre-Obadia N, Antal A, Ayache SS, Baeken C, Benninger DH, Cantello RM, Cincotta M, de Carvalho M, De Ridder D, Devanne H, Di Lazzaro V, Filipovic SR, Hummel FC, Jaaskelainen SK, Kimiskidis VK, Koch G, Langguth B, Nyffeler T, Oliviero A, Padberg F, Poulet E, Rossi S, Rossini PM, Rothwell JC, Schonfeldt-Lecuona C, Siebner HR, Slotema CW, Stagg CJ, Valls-Sole J, Ziemann U, Paulus W, Garcia-Larrea L. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS). Clin Neurophysiol. 2014 Nov;125(11):2150-2206. doi: 10.1016/j.clinph.2014.05.021. Epub 2014 Jun 5. PMID 25034472
- [Background] Stultz DJ, Osburn S, Burns T, Pawlowska-Wajswol S, Walton R. Transcranial Magnetic Stimulation (TMS) Safety with Respect to Seizures: A Literature Review. Neuropsychiatr Dis Treat. 2020 Dec 7;16:2989-3000. doi: 10.2147/NDT.S276635. eCollection 2020. PMID 33324060
- [Background] Lerner AJ, Wassermann EM, Tamir DI. Seizures from transcranial magnetic stimulation 2012-2016: Results of a survey of active laboratories and clinics. Clin Neurophysiol. 2019 Aug;130(8):1409-1416. doi: 10.1016/j.clinph.2019.03.016. Epub 2019 Apr 6. PMID 31104898